CLINICAL TRIAL: NCT05245760
Title: ChemoRadiation And Tislelizumab for Esophageal/EGJ Cancer
Acronym: CRATER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable.
Sponsor: Zhonglin Hao (Other)
Collaborators: BeiGene (Industry); University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Zhonglin Hao, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21-LUN-125-PMC
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Cancer; Esophagogastric Junction Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Immunotherapy; Drug Therapy; Carboplatin; Paclitaxel; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patient (Experimental): All patients receive Tislelizumab, q3week; chemotherapy with carboplatin and paclitaxel weekly concurrently for 5 weeks before surgery. Tislelizumab is continued q3week in all patients after surgery for a total of one year from the start of study.
  Interventions: Drug: Intravenous Tislelizumab; Drug: Chemotherapy; Radiation: Fractionated radiation; Procedure: Esophagectomy

INTERVENTIONS:
Drug: Intravenous Tislelizumab — Participants will receive 200mg, every three weeks for up to 51 weeks
  Other Names: immunotherapy
Drug: Chemotherapy — Carboplatin (AUC2) and Paclitaxel (50mg/m2), Weekly x 5 weeks
  Other Names: carboplatin and paclitaxel
Radiation: Fractionated radiation — Concurrent with chemo, x5 weeks
Procedure: Esophagectomy — Surgical resection of cancer after chemoradiation therapy when no disease progression found.

SUMMARY:
This study aims to determine the effects of chemoradiation and Tislelizumab on Esophageal/EGJ Cancer before and after surgery.

DETAILED DESCRIPTION:
Esophageal cancer patients in this trial will receive chemoradiation therapy with tislelizumab, which is an anti-PD-1 antibody, before surgery. Patient will be evaluated for complete pathological response or major pathological response rate following chemoradiation. Patient will continue on to get tislelizumab after surgery to complete total of a year of treatment. They will be evaluated for PFS and OS. Throughout the study, drug tolerability and toxicities will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments
2. Age ≥ 18 years but 80 years or younger on the day of signing the informed consent form.
3. Histologically proven esophageal squamous cell cancer or adenocarcinoma.
4. De novo diagnosis, have not received prior treatment
5. AJCC 8. T1N1 or T2-4aN0-2M0 resectable disease
6. ECOG Performance Status ≤ 1
7. Adequate organ function as indicated by the following laboratory values

   a. Patients must not have required a blood transfusion or growth factor support ≤ 14 days before sample collection at screening for the following i. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L ii. Platelets ≥ 100 x 109/L iii. Hemoglobin ≥ 90 g/L b. Serum creatinine ≤ 1.5 x ULN (upper limit of normal) or estimated Glomerular Filtration Rate ≥ 60 mL/min/1.73 m2 c. Serum total bilirubin ≤ 1.5 x ULN (total bilirubin must be < 3 x ULN for patients with Gilberts syndrome). d. AST and ALT ≤ 3 x ULN
8. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥ 120 days after the last dose of tislelizumab, and have a negative urine or serum pregnancy test ≤ 7 days before the first dose of tislelizumab.
9. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of tislelizumab

   Exclusion Criteria:
10. Unresectable disease either T4b or M1 per AJCC8
11. Deemed inoperable for any reason by attending surgeon
12. Any prior treatment directed at the tumor except biopsy.
13. Active autoimmune diseases such as SLE, RA requiring systemic immunosuppression or history of autoimmune diseases that may relapse.
14. Any active malignancy ≤ 2 years before first dose of study drug, except for cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast)
15. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before tislelizumab. Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:

    1. Adrenal replacement steroid (dose ≤ 15 mg daily of prednisone or equivalent)
    2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
    3. Short course (≤ 7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)
16. Laboratory test abnormalities in potassium, sodium, or corrected calcium > Grade 1 despite standard medical management
17. History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
18. Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc.
19. A known history of HIV infection not controlled with anti-retroviral therapy
20. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is > 500 IU/mL or patients with active hepatitis C virus (HCV) should be excluded. Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA < 500 IU/mL), and cured hepatitis C patients can be enrolled
21. Prior allogeneic stem cell transplantation or organ transplantation
22. Any of the following cardiovascular risk factors:

    1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before first dose of tislelizumab and chemotherapy
    2. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV (Appendix 6) ≤ 6 months
    3. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months prior to initiation of treatment on study.
23. A history of severe hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
24. Has received radiation therapy within 4 weeks, chemotherapy, immunotherapy (e.g., interleukin, interferon, thymosin), or any investigational therapies within 14 days or 5 half lives (whichever is shorter) of the first study drug administration
25. Was administered a live vaccine ≤ 4 weeks before tislelizumab Note: Seasonal vaccines for influenza are generally inactivated vaccines and are allowed.

    Intranasal vaccines are live vaccines and are not allowed. The mRNA vaccine for SARSCoV2 is allowed if the second dose is administered two weeks before study drug is administered.
26. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that, will be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct.
27. Concurrent participation in another therapeutic clinical study.
28. History of allergy to platinum or taxane
29. Li-Fraumeni Syndrome where radiation is contraindicated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | 12 months
  Pathological complete response (pCR) rate in patients treated with tislelizumab and chemoradiation followed by surgery. The pCR rate will be estimated by number of patients who has had pCR divided by the total number of evaluable patients treated with neoadjuvant therapy before surgery. The exact 95% confidence interval of the pCR rate will be provided.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 12 months
  The time from the participants' date of surgery to the date of disease progression or death, whichever occurs first
Major pathological response (MPR) | 12 months
  The number of patients who had 90% or more tumor showing necrosis divided by the total number of evaluable patients treated with neoadjuvant therapy before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhonglin Hao, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No